CLINICAL TRIAL: NCT03430973
Title: Driving Simulation Experiments of Aggressive Driving and Road Rage
Brief Title: Aggressive Driving and Road Rage: A Driving Simulation Experiment.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Thomas Kerwin, Director of Operations OSU Driving Simulation Lab, Ohio State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 2018B0081
Record Dates: First submitted 2018-01-23; First posted 2018-02-13 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Aggression
Keywords: aggressive driving; road rage
MeSH Terms: conditions — Aggression; Road Rage | interventions — Videotape Recording; Ethanol; Music Therapy

STUDY DESIGN:
Intervention Model Description: Seven driving simulation experiments on aggressive driving and road rage (see descriptions above).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Experiment 1 (Experimental): The purpose of Experiment 1 is to develop a standardized measure of aggressive driving for driver simulation experiments. After giving their consent, participants (N=200) will complete several personal variables (i.e., gender, age, driving experience, driving frequency, trait anger, self-reported aggressive and prosocial driving). Next, participants will watch several short videos of aggressive driving (e.g., speeding, tailgating, driving on shoulder), and road rage (e.g., hitting another vehicle or pedestrian). Participants will indicate whether the driver's behavior was aggressive (yes, no), and will rate how aggressive it was on an 11-point scale (0=not at all aggressive to 10=extremely aggressive). A debriefing will follow.
  Interventions: Behavioral: Videos
- Experiment 2 (Experimental): Experiment 2 tests whether participants actually drive more aggressively after a playing a violent or nonviolent racing video game. After giving their consent, participants (N=60, n=30 each group) will complete the same personal variables as in Experiment 1, and will report the video games they play. Next, participants will be randomly assigned to play one of two types of video games for 20 minutes: (1) violent racing video game, (2) nonviolent racing game, or (3) a neutral game. After participants complete the driving scenario, participants will complete measures of state and hostile appraisals. A debriefing will follow.
  Interventions: Behavioral: Video game
- Experiment 3 (Experimental): Experiment 3 tests the effects of racial bumper stickers on black and white participants. After giving their consent, participants (N=120; n=60 black, n=60 white) will complete the personal variables (see Experiment 1), the race IAT, and report their political party. Some cars in the driving scenario will contain bumper stickers. Experiment 3 contains four conditions: (1) white participants / "All Lives Matter" stickers, (2) black participants / "All Lives Matter" stickers, (3) white participants / "Black Lives Matter" stickers, (4) black participants / "Black Lives Matter" stickers. After participants complete the driving scenario, they will complete measures of state and hostile appraisals, and will report their attitudes toward the #BLM and #ALM movements. A debriefing will follow.
  Interventions: Behavioral: Bumper stickers
- Experiment 4 (Experimental): Experiment 4 tests the effects of political bumper stickers on aggressive driving in Republicans versus Democrats. After giving their consent, participants (N=120; n=60 Republicans, n=60 Democrats) will complete the personal variables (see Experiment 1). Some cars in the driving scenario will contain bumper stickers. Experiment 4 has four conditions: (1) Republicans / "Donald Trump for President 2016" stickers, (2) Republicans / "Hillary Clinton for President 2016" stickers, (3) Democrats / "Donald Trump for President 2016" stickers, (4) Democrats / "Hillary Clinton for President 2016" stickers. After participants complete the driving scenario, they will complete measures of state and hostile appraisals, and will report their attitudes toward Trump and Clinton. A debriefing will follow.
  Interventions: Behavioral: Bumper stickers
- Experiment 5 (Experimental): Experiment 5 tests whether alcohol-related cues can increase aggressive driving. After giving their consent, participants (N=40) will complete the personal variables (see Experiment 1). Next, participants will be randomly assigned to one of two conditions: (1) 12-pack of beer on passenger seat, or (2) 12-pack of sparkling water on passenger seat. Participants will be told that the object on the seat is part of a different experiment that the other experimenter forgot to clean up, which they should ignore it. After participants complete the driving scenario, they will complete measures of state and hostile appraisals, and will be debriefed.
  Interventions: Behavioral: Alcohol-related cues
- Experiment 6 (Experimental): Experiment 6 will test the effects of music with aggressive versus prosocial lyrics on aggressive driving. The tempo of the music will also be manipulated because it might influence arousal levels. After giving their consent, participants (N=150, n=30 per group) will complete the personal variables (see Experiment 1). Music will be played over the car's sound system. Participants will be randomly assigned to one of five conditions: (1) violent lyrics / upbeat tempo, (2) violent lyrics / calm tempo, (3) prosocial lyrics / upbeat tempo, (4) prosocial lyrics / calm tempo, or (5) no music control. After participants complete the driving scenario, they will complete measures of state and hostile appraisals, and will be debriefed.
  Interventions: Behavioral: Music
- Experiment 7 (Experimental): Experiment 7 tests whether roadside vegetation can reduce aggression in frustrated drivers. After giving their consent, participants (N=90, n=30 per group) will complete the personality variables (see Experiment 1). Next, they will complete the Enjoyment of Nature Scale (Cheng & Moore, 2012), which contains 7 items (e.g., "I like to see wild flowers in nature" and "Being in the natural environment makes me feel peaceful"; 1=strongly disagree to 5= strongly disagree; Cronbach =.87). Next, participants will be randomly assigned to one of three driving scenarios: (1) roadside vegetation, (2) trash, or (3) control (no roadside vegetation / no trash). After participants complete the driving scenario, they will complete measures of state and hostile appraisals, and will be debriefed.
  Interventions: Behavioral: Roadside vegetation

INTERVENTIONS:
Behavioral: Videos — Videos depicting various aggressive driving and road rage behaviors.
  Arms: Experiment 1
Behavioral: Bumper stickers — Bumper stickers hypothesized to increase or decrease aggressive driving.
  Arms: Experiment 3; Experiment 4
Behavioral: Alcohol-related cues — Case of beer or water on passenger seat.
  Other Names: beer water
  Arms: Experiment 5
Behavioral: Music — Lyrics and tempo of music will be manipulated to increase or decrease aggressive driving.
  Arms: Experiment 6
Behavioral: Roadside vegetation — The roadside will contain trash to increase aggressive driving, or vegetation to decrease aggressive driving. There is also a control group.
  Arms: Experiment 7
Behavioral: Video game — Participants will play a racing or neutral video game before driving in the simulator.
  Arms: Experiment 2

SUMMARY:
Driving a car is the most dangerous behavior most people engage in every day. According to the World Health Organization, about 1.25 million people die each year as a result of road traffic crashes, and they are the leading cause of death among 15 to 29 year olds. According to the National Highway Traffic Safety Administration, 37,461 Americans were killed in motor vehicle crashes in 2016 - about 103 per day. Although there are several causes of traffic crashes (e.g., texting, alcohol consumption, inclement weather), the leading cause is aggressive driving. In the United States, aggressive driving accounts for more than half of all traffic fatalities. Thus, aggressive driving is an important applied health topic, especially for young drivers.

DETAILED DESCRIPTION:
Experimental studies are needed to draw inferences about the causes of aggressive driving. Only six driving simulation experiments have been conducted, and one of these experiment was conducted by the investigators (Bushman, Kerwin, Whitlock, & Weisenberger, 2017).

The proposed research will test the effects of seven situational risk factors: (1) racing video games (Experiment 2), (2) racial bumper stickers (i.e., "Black Lives Matter" bumper stickers for white motorists vs. "All Lives Matter" bumper stickers for black motorists; Experiment 3), (3) political bumper stickers (i.e., "Donald Trump for President 2016" for Democrat motorists vs. "Hillary Clinton for President 2016" for Republican motorists; Experiment 4), (4) alcohol-related cues (i.e., a case of beer vs. water on the passenger seat; Experiment 5), (5) music with violent lyrics (Experiment 6), (6) music with an upbeat tempo (Experiment 6), and (7) roadside trash (Experiment 7). The proposed research will also test the effects of five situational protective factors: (1) racial bumper stickers (i.e., "Black Lives Matter" for black motorists vs. "All Lives Matter" for white motorists; Experiment 3), (2) political bumper stickers (i.e., "Donald Trump for President 2016" for Republican motorists vs. "Hillary Clinton for President 2016" for Democrat motorists; Experiment 4), (3) music with prosocial lyrics (Experiment 6), (4) music with a calm tempo (Experiment 6), and (5) roadside vegetation (Experiment 7).

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adults recruited from Central Ohio (Franklin County) through advertisements (e.g., newspaper, Internet).
* Participants' ages will vary depending on the experiment. 18 and older for Experiment 1; 18-21 for Experiments 2-4 and 6-7; 21+ for Experiment 5
* All participants must have a current driver license.

Exclusion Criteria:

• Participants who have motion sickness will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Aggressive driving behavior | Observed in driving scenario during the experimental session
  The two primary measures of aggressive driving will be tailgating and speeding. Tailgating measures are based on the number of seconds between the participant's car and the car in front of them: (1) 4-second rule (recommended for speeds above 30 MPH, in heavy traffic, or when there are many obstacles, as in the present driving scenario), (2) 3-second rule (dangerous), and (3) 2-second rule (extremely dangerous). Average speed is a poor measure of speeding because it depends heavily on random influences. Instead, a relatively high-speed cutoff (e.g., 50 MPH) will be used before averaging because it removes the variability due to traffic. Other measures of aggressive driving include off-road driving (e.g., crossing the double solid yellow lines into oncoming traffic, driving on the shoulder), horn honking, verbal aggression, and aggressive gestures (e.g., giving another driver the middle finger). Measures of aggressive driving will be combined to reduce Type I errors.
Road rage | Observed in driving scenario during the experimental session, up to one hour.
  The four primary measures of road rage will be colliding into other vehicles, motorcyclists, bicyclists, and pedestrians. Acts of road rage are expected to occur far less frequently than acts of aggressive driving. Acts of road rage will be combined to reduce Type I errors.

SECONDARY OUTCOMES:
State anger | Immediately after completing driving scenario, during the experimental session, up to one hour.
  In the proposed research, state anger will be measured using the State Anger Scale (Spielberger, 1988), which contains 15 items (e.g., "I feel angry") that are rated on a 4-point scale (1 = Not at all; 2 = Somewhat; 3 = Moderately so; 4 = Very much so; Cronbach = .93).
Hostile attributions | Immediately after completing driving scenario, during the experimental session, up to one hour.
  Research has shown that the hostile attribution bias can influence appraisal and decision processes. The hostile attribution bias is the tendency to perceive ambiguous actions by others as aggressive. For example, if a driver cuts you off, a hostile attribution would be that the driver did it purposely (not accidentally). Research has shown that attributing causality to an offending driver predicts aggressive driving. In the proposed research, we will measure whether people assign blame to other drivers using a measure successfully used in previous research. For each provocative event, participants will be asked whether the actions of the other driver were intentional or accidental. For example, "Do you think the other driver deliberately cut you off?" vs. "I think the other driver cut me off by accident" (1=Not at all to 7=Very much so). In Experiments 2-4, 6-7, we expect hostile appraisals to be positively related to aggressive driving. This measure is not included in Experiment 5.

OTHER OUTCOMES:
Trait anger | Completed after consent is signed, before the driving simulation experiment begins.
  Trait anger is a personality dimension that reflects the person's chronic tendency to experience the emotion of state anger with greater frequency, intensity, and duration. Trait anger is an important antecedent of state anger and aggression. Trait anger will be measured using the Trait Anger Scale, which contains 10 items (e.g., "I have a fiery temper") that are rated on a 4-point scale (1 = Almost never; 2 = Sometimes; 3 = Often; 4 = Almost always)
Narcissism | Completed after consent is signed, before the driving simulation experiment begins.
  Narcissism is characterized by excessive self-love and a selfish orientation. Previous research has shown that narcissism is a risk factor for aggressive driving.
  Narcissism will be measured using the Single Item Narcissism Scale (SINS): "To what extent do you agree with this statement: 'I am a narcissist.' (Note: The word "narcissist" means egotistical, self-focused, vain, etc.)," which is scored using a 7-point scale (1 = Not very true of me to 7 = Very true of me).
Empathy | Completed after consent is signed, before the driving simulation experiment begins.
  Empathy involves feeling compassion for others and imagining how they feel. We expect empathy to be negatively related to aggressive driving. Empathy will be measured using the Single Item Trait Empathy Scale (SITES): "To what extent does the following statement describe you: 'I am an empathetic person.' (Note: An empathetic person understands others' feelings, and experiences care and concern for them.)," which is scored using a 5-point scale (Not very true of me to 5 = Very true of me)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Bushman, PhD, Study Director — Ohio State University
Locations (1):
- The Ohio State University Driving Simulation Laboratory, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data set and syntax will be posted to figshare.com
Supporting Information: Analytic Code
Time Frame: After an experiment is accepted for publication, the data will be uploaded with no time limit.
Access Criteria: The data will be posted on an open access webpage - figshare
URL: https://figshare.com

REFERENCES:
- [Background] Bushman, B. J., Kerwin, T., Whitlock, T., & Weisenberger, J. M. (2017). The weapons effect on wheels: Motorists drive more aggressively when there is a gun in the vehicle. Journal of Experimental Social Psychology, 73, 82-85. doi:10.1016/j.jesp.2017.06.007
- [Background] Cheng, J. C., & Monroe, M. C. (2012). Connection to nature: Children's affective attitude toward nature. Environment and Behavior, 44(1), 31-49. doi:10.1177/0013916510385082
- [Background] Spielberger, C. D. (1988). State-trait anger expression inventory: STAXI professional manual. Odessa, FL: Psychological Assessment Resources.
- [Background] Wickens CM, Wiesenthal DL, Flora DB, Flett GL. Understanding driver anger and aggression: attributional theory in the driving environment. J Exp Psychol Appl. 2011 Dec;17(4):354-70. doi: 10.1037/a0025815. Epub 2011 Oct 10. PMID 21988326

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Experiment 2 adjusted (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT03430973/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: Experiment 5 adjusted (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT03430973/Prot_SAP_000.pdf